CLINICAL TRIAL: NCT01249443
Title: A Phase 1 Study of Paclitaxel and Carboplatin in Solid Tumors (With Focus on Upper Aerodigestive Cancers) in Persons With HIV Infection
Brief Title: Paclitaxel and Carboplatin in Treating Patients With Metastatic or Recurrent Solid Tumors and HIV Infection
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Inadequate accrual rate
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); The Emmes Company, LLC (Industry); University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC-078; NCI-2011-02511 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000689900 (Registry Identifier: clinicaltrials.gov); AMC-078 (Other: AIDS - Associated Malignancies Clinical Trials Consortium); AMC-078 (Other: CTEP); U01CA121947 (NIH)
Record Dates: First submitted 2010-11-25; First posted 2010-11-29 (Estimated); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: HIV Infection; Recurrent Anal Cancer; Recurrent Breast Cancer; Recurrent Esophageal Cancer; Recurrent Gastric Cancer; Recurrent Metastatic Squamous Neck Cancer With Occult Primary; Recurrent Non-small Cell Lung Cancer; Recurrent Ovarian Epithelial Cancer; Recurrent Salivary Gland Cancer; Recurrent Squamous Cell Carcinoma of the Hypopharynx; Recurrent Squamous Cell Carcinoma of the Larynx; Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Squamous Cell Carcinoma of the Nasopharynx; Recurrent Squamous Cell Carcinoma of the Oropharynx; Recurrent Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Recurrent Verrucous Carcinoma of the Larynx; Recurrent Verrucous Carcinoma of the Oral Cavity; Salivary Gland Squamous Cell Carcinoma; Stage IV Anal Cancer; Stage IV Breast Cancer; Stage IV Esophageal Cancer; Stage IV Gastric Cancer; Stage IV Non-small Cell Lung Cancer; Stage IV Ovarian Epithelial Cancer; Stage IV Salivary Gland Cancer; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Larynx; Stage IV Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IV Squamous Cell Carcinoma of the Nasopharynx; Stage IV Squamous Cell Carcinoma of the Oropharynx; Stage IV Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IV Verrucous Carcinoma of the Larynx; Stage IV Verrucous Carcinoma of the Oral Cavity; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — HIV Infections; Anus Neoplasms; Breast Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Ovarian Epithelial; Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Vorinostat; Carboplatin; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (carboplatin, paclitaxel) (Experimental): Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 3. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Before February 1, 2013, patients also received vorinostat PO once daily on days 1-5 with paclitaxel and carboplatin.
  Interventions: Drug: vorinostat; Other: diagnostic laboratory biomarker analysis; Other: pharmacological study; Drug: carboplatin; Drug: paclitaxel

INTERVENTIONS:
Drug: vorinostat — Given PO
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
Other: diagnostic laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol

SUMMARY:
This phase I clinical trial is studying the side effects and the best dose of vorinostat when given together with paclitaxel and carboplatin in treating patients with metastatic or recurrent solid tumors and human immunodeficiency virus (HIV) infection. Vorinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving vorinostat together with paclitaxel and carboplatin may kill more tumor cells.

NOTE: An administrative decision was made by NCI to halt further study of vorinostat in this specific patient population as of February 1, 2013. No patients remain on vorinostat. Going forward this study will determine the safety and tolerability of the paclitaxel and carboplatin combination in this patient population.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability of vorinostat in combination with paclitaxel and carboplatin in solid tumor patients with HIV infection.

II. To determine the maximal tolerated dose (MTD) of the combination in this patient population.

*NOTE: An administrative decision was made by Cancer Therapy Evaluation Program (CTEP) to halt further study of vorinostat in this specific patient population as of February 1, 2013, and no patients remain on vorinostat. The primary objective going forward will determine the safety and tolerability of the paclitaxel and carboplatin combination in this patient population.

SECONDARY OBJECTIVES:

I. To preliminarily assess response rates of the therapeutic combination in lung, head and neck, and esophageal cancers.

II. To evaluate the pathological characteristics of non-acquired immunodeficiency syndrome (AIDS) defining cancers of the upper aerodigestive tract.

III. To determine the presence and oncogenic activity of human papillomavirus (HPV) infection in tumor tissues and to correlate HPV infection with clinical outcomes.

IV. To investigate possible pharmacokinetic interactions between paclitaxel and antiretroviral therapy in persons with HIV infection.

OUTLINE: This is a multicenter, dose-escalation study of vorinostat followed by an expansion cohort study.

Patients receive vorinostat orally (PO) once daily on days 1-5 and paclitaxel intravenously (IV) over 3 hours and carboplatin IV over 30 minutes on day 3. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Some patients undergo blood sample collection at baseline and periodically during course 1 for pharmacokinetic studies and HIV viral load analysis.

Note: An administrative decision was made by CTEP to halt further study of vorinostat in this specific patient population as of February 1, 2013. No patients remain on vorinostat. The primary objective going forward will determine the safety and tolerability of the paclitaxel and carboplatin combination in this patient population, without vorinostat. The information pertaining to vorinostat is for historical purposes.

After completion of study therapy, patients are followed up every 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have known HIV infection and histologically confirmed solid malignancy that is metastatic or unresectable and is therefore incurable; although the focus of this trial will be on upper aerodigestive cancers (non-small cell lung cancer, head and neck squamous cell carcinoma, and non-gastroesophageal junction esophageal cancer), patients with other incurable solid tumor with disease potentially sensitive to carboplatin and/or taxanes (including but not limited to salivary gland cancer, gastric cancer, breast cancer, ovarian cancer, or anal cancer, BUT excluding Kaposi sarcoma), will be eligible
* Up to 1 prior systemic therapy regimen will be permitted for palliative treatment of metastatic or unresectable relapsed disease; however, previous chemotherapy delivered with curative-intent (i.e., chemoradiotherapy or adjuvant [postoperative] chemotherapy at a time disease was considered potentially curable) will be permitted; prior taxane (including paclitaxel or docetaxel) and/or platinum exposure will be permitted; however, patients must not experience disease progression within 3 months of platinum-based therapy; at least 4 weeks must have elapsed since prior chemotherapy or radiation therapy, 6 weeks if the last regimen included carmustine (BCNU) or mitomycin C; toxicities from prior anticancer therapy must have recovered to =< Grade 1
* Serologic documentation of HIV infection at any time prior to study entry, as evidenced by positive enzyme-linked immunosorbent assay (ELISA), positive Western Blot, or any other federally approved licensed HIV test; a positive HIV viral load prior to study entry will also be permitted
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 50%)
* Documented life expectancy of greater than 12 weeks
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST)(serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamic-pyruvic transaminase [SGPT]) =< 2.5 X institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 50 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Additionally, serum magnesium and potassium must be within institutional normal limits, and a CD4 count > 100/mcL will be required within 2 weeks of study participation
* Presence of at least one measureable tumor lesion is required
* Participating patients must receive medically appropriate care and treatment for HIV infection, including antiretroviral medications, when clinically indicated, and should be under the care of a physician experienced in HIV management; with the exception of treatment with zidovudine and stavudine, patients will be eligible regardless of antiretroviral regimen (no antiretroviral therapy, nonnucleoside reverse transcriptase inhibitors [NNRTI]-based therapy, or protease inhibitor based therapy), provided there is no intention to initiate therapy or the regimen has been stable for at least 4 weeks with no intention to change the regimen within 8 weeks following study entry; the exact regimen used for HIV therapy will be captured on Case Report Forms; as study-specific (antiretroviral therapy-based) strata fill, however, only patients fitting the remaining open strata will be accrued
* Because histone deacetylase inhibitors as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, during the duration of study participation, and for at least 3 months following study completion; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately; women of child-bearing potential must have a negative pregnancy test within 7 days before initiation of study drug dosing; post menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential; (Note: A woman of childbearing potential is one who is biologically capable of becoming pregnant; this includes women who are using contraceptives or whose sexual partners are either sterile or using contraceptives)
* Ability to understand and the willingness to sign a written informed consent document; as the correlative studies are critical to the clinical and scientific value of the trial, CD4 count/HIV viral load determinations will be required, and participation in the tumor-based correlative studies will be strongly recommended; additionally, investigators MUST request sample donation to the AIDS Cancer Specimen Resource (ACSR); however, the patient may refuse sample donation; patients accrued to the expansion phase of the study will be required to undergo pharmacokinetic sampling
* Subjects must in the opinion of the Investigator be capable of complying with this protocol

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events (toxicities not improved to =< Grade 1) due to agents administered more than 4 weeks earlier; additionally, patients experiencing disease progression within 3 months of platinum-based therapy will be excluded from trial participation
* Due to availability of effective first- and second-line therapies (as well as disease-specific clinical trials), patients with diagnosis of active Kaposi sarcoma will be excluded from study participation; however, persons with other active malignancy with prior history of Kaposi sarcoma can be considered for participation at the discretion of the Study Chair
* Patients may not be receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to the study agents used in study (including hypersensitivity to paclitaxel, Cremophor, or platins)
* For subjects assigned to take vorinostat, inability to take oral medications; vorinostat capsules must be administered whole; note: this criterion does NOT apply to subjects treated on the Expansion Cohort (accruals post February 1, 2013)
* As ketoconazole may inhibit paclitaxel metabolism, patients receiving ketoconazole for any treatment indication are ineligible; patients receiving any other medications or substances that are inhibitors or inducers of CYP450 enzymes will be eligible; however, use all such medications or substances must be documented in the Case Report Forms
* For subjects assigned to take vorinostat, prior exposure to vorinostat or other known histone deacetylase (HDAC) inhibitors for cancer therapy; patients should not have taken valproic acid, another histone deacetylase inhibitor, for at least 2 weeks prior to study enrollment; note: this criterion does NOT apply to subjects treated on the Expansion Cohort (accruals post February 1, 2013)
* Since zidovudine and stavudine have potential for severe hematological toxicity potentially overlapping with toxicities of the study therapy, treatment with these agents will be disallowed
* Due to potential toxicity associated with study therapy (particularly with paclitaxel), patients with peripheral neuropathy > Grade 1 will be excluded from study participation
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, opportunistic infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements; patients with HIV infection will be eligible provided they meet the criteria specified; patients with known Hepatitis B infection should be screened for active disease prior to study participation; patients with chronic Hepatitis C infection will be eligible at the discretion of the treating investigator
* Pregnant women are excluded from this study and women who become pregnant while on study must be immediately discontinued; women who are breastfeeding will not be eligible for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events during paclitaxel and carboplatin treatment according to dose-limiting toxicities (DLTs), graded using Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0) | 21 days

SECONDARY OUTCOMES:
Response rates in patients with lung, head and neck, and esophageal cancers assessed by Response Evaluation Criteria for Solid Tumors (RECIST) 1.1 | Up to 3 years
  For each stratum, binomial proportions and their 95% confidence intervals will be used to preliminarily assess response rates of the therapeutic combination in lung, head and neck, and esophageal cancers.
Effects of therapy on HIV viral load and CD4 cell count | Baseline and at 6, 12, and 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Missak Haigentz, Principal Investigator — AIDS Associated Malignancies Clinical Trials Consortium
Locations (10):
- United States (10):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UCLA Center for Clinical AIDS Research and Education, Los Angeles, California
  - Lombardi Comprehensive Cancer Center at Georgetown University, Washington D.C., District of Columbia
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - John H. Stroger Jr. Hospital of Cook County, Chicago, Illinois
  - Boston Medical Center, Boston, Massachusetts
  - Siteman Cancer Center at Washington University, St Louis, Missouri
  - Montefiore Medical Center, The Bronx, New York
  - Pennsylvania Oncology Hematology Associates, Philadelphia, Pennsylvania
  - Benaroya Research Institute at Virginia Mason, Seattle, Washington

REFERENCES:
- [Derived] Haigentz M, Moore P, Bimali M, Cooley T, Sparano J, Rudek M, Ratner L, Henry D, Ramos J, Deeken J, Rubinstein P, Chiao E. Safety and Tolerability of Carboplatin and Paclitaxel in Cancer Patients with HIV (AMC-078), an AIDS Malignancy Consortium (AMC) Study. Oncologist. 2022 Aug 5;27(8):623-e624. doi: 10.1093/oncolo/oyac004. PMID 35429391